CLINICAL TRIAL: NCT00139997
Title: A Multicenter, Randomized Controlled Trial of Negative Ion Generation Versus Light-Emitting Diode Phototherapy For Seasonal Affective Disorder
Brief Title: Environmental Treatment for Seasonal Affective Disorder (SAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University Medical Center Groningen (Other); University of British Columbia (Other); Royal Ottawa Mental Health Centre (Unknown); Douglas Hospital Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22,777; 22,777 (Other: Yale University)
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-01

CONDITIONS: Seasonal Affective Disorder
Keywords: Major Depression; Seasonal Affective Disorder (SAD)
MeSH Terms: conditions — Seasonal Affective Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LED phototherapy device (Experimental): Litebook treatment devices: LED phototherapy device, used for 30 min before 8 am
  Interventions: Device: Litebook treatment devices
- Inactivated Negative Ion Generator (Placebo Comparator): Equivalent exposure to inactivated negative ion generator
  Interventions: Device: Inactivated negative ion generator

INTERVENTIONS:
Device: Litebook treatment devices — Litebook LED phototherapy device used for 30 min before 8 am
  Arms: LED phototherapy device
Device: Inactivated negative ion generator — Equivalent exposure to inactivated negative ion generator
  Arms: Inactivated Negative Ion Generator

SUMMARY:
The purpose is to study treatments of Seasonal Affective Disorder (SAD).

DETAILED DESCRIPTION:
This is a multicenter, randomized controlled trial of negative ion generation versus light-emitting diode phototherapy for seasonal affective disorder. Participants appropriate for the study are subjects with a DSM IV diagnosis of Major Depression, with seasonal pattern, winter type. Subjects were seen at Yale University,New Haven,CT University of British Columbia,Vancouver,BC Groningen University Hospital,Groningen, The Netherlands, Royal Ottawa Hospital, Ottawa,Ontario, McGill University, Montreal,Quebec, University Hospital,Saskatoon, Saskatchewan. The trial is 4 weeks in duration.

This trial has now been completed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet DSM-IV criteria for major depressive episodes with a seasonal pattern, winter type.

Exclusion Criteria:

* Significant suicidal risk
* Serious medical illness
* Pregnancy
* Other DSM-IV diagnoses
* Taking mood altering medication
* May not travel to a sunny destination during study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul H. Desan, PhD, MD, Principal Investigator — Yale New Haven Hospital
Locations (5):
- Yale University School of Medicine, New Haven, Connecticut, United States
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Royal Ottawa Mental Health Centre, , Ontario, K1Z 7K4 Canada, Ottawa, Ontario
  - Douglas Hospital Research Centre, Montreal, Quebec
- University Medical Center Groningen, Groningen, RB, Netherlands

REFERENCES:
- [Result] Desan PH, Weinstein AJ, Michalak EE, Tam EM, Meesters Y, Ruiter MJ, Horn E, Telner J, Iskandar H, Boivin DB, Lam RW. A controlled trial of the Litebook light-emitting diode (LED) light therapy device for treatment of Seasonal Affective Disorder (SAD). BMC Psychiatry. 2007 Aug 7;7:38. doi: 10.1186/1471-244X-7-38. PMID 17683643

RESULTS

PARTICIPANT FLOW:
Groups:
- LED Phototherapy: Phototherapy with light-emitting diode phototherapy device
- Inactive Intervention: Equivalent exposure to inactive negative ion generator
Period: Overall Study
Arm/Group | LED Phototherapy | Inactive Intervention
Started | 15 | 11
Completed | 14 | 9
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LED Phototherapy | Inactive Intervention | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.4) | 44.9 (10.4) | 43.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
  Canada | 6 | 3 | 9
  Netherlands | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage SIGH SAD (Structured Interview Guide For The Hamilton Depression Rating Scale), SAD Version
Description: SIGH SAD Structured Interview Guide for the Hamilton Depression Rating Scale, Seasonal Affective Disorder (SAD)version. The items are augmented with additional items to reflect better the atypical depressive symptoms usually seen in SAD, eg, increased sleep, weight, appetite and fatigue. On this scale, higher scores reflect increased depression intensity. The maximum score attainable is 63, and the minimum is 0. A score of less than 9 is regarded as consistent with normal mood, the absence of major depression.
  Calculated: SIGH SAD score at trial end x 100 / SIGH SAD score at randomization
Time Frame: Week 4
Population: These participants are analyzed ITT- last observation carried forward.
Measure: Mean (Standard Deviation); unit: Percentage of SIGH SAD
Arm/Group | LED Phototherapy | Inactive Intervention
Number analyzed (Participants) | 15 | 11
Percentage of SIGH SAD | 34.5 (30.47) | 60.4 (23.61)
Statistical Analysis 1: Comparison: LED Phototherapy vs Inactive Intervention; Test type: Superiority or Other; p = 0.028, t-test, 2 sided

2. Secondary Outcome: SIGH SAD (Structured Interview Guide For The Hamilton Depression Rating Scale), SAD Version
Description: SIGH SAD Structured Interview Guide for the Hamilton Depression Rating Scale, SIGH SAD Structured Interview Guide for the Hamilton Depression Rating Scale, Seasonal Affective Disorder (SAD)version. This is a structured interview, which is an interview in which the clinician is provided exact questions to use to inquire about symptoms of depression and explicit standards for rating the intensity of each symptom item. The interview assesses the symptoms which make up the Hamilton Depression Rating Scale, which is the standard in the majority of clinical trials in depression. The items are augmented with additional items to reflect better the atypical depressive symptoms usually seen in SAD, eg, increased sleep, weight, appetite and fatigue. On this scale, higher scores reflect increased depression intensity. The maximum score attainable is 63, and the minimum is 0. A score of less than 9 is regarded as consistent with normal mood, the absence of major depression.
Time Frame: Weekly following randomization
Population: These participants are analyzed ITT- last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LED Phototherapy | Inactive Intervention
Number analyzed (Participants) | 15 | 11
units on a scale
  Randomization | 28.0 (5.3) | 25.1 (3.2)
  Week 1 | 18.6 (7.9) | 19.0 (7.2)
  Week 2 | 14.9 (10.0) | 17.9 (4.9)
  Week 3 | 11.1 (10.1) | 14.9 (4.2)
  Week 4 | 8.7 (8.4) | 13.4 (5.4)

ADVERSE EVENTS:
Arm/Group | LED Phototherapy | Inactive Intervention
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 2/15 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LED Phototherapy (N=15) | Inactive Intervention (N=11)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
dry mouth (General disorders) | 1 (1) | 0 (0)
jitteriness (Psychiatric disorders) | 1 (1) | 1 (1)
difficulty falling asleep (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No